CLINICAL TRIAL: NCT01874704
Title: Comparison of Biomarkers of Stress in Emergency Physicians Working a 24-hour Shift or a 14-hour Night Shift - the JOBSTRESS Randomized Trial
Acronym: JOBSTRESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: Association des Médecins des Urgences de Clermont-Ferrand (Other); Université d'Auvergne (Other)
Responsible Party: Sponsor
Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: CHU-0154; 2009-A01309-48
Record Dates: First submitted 2013-05-24; First posted 2013-06-11 (Estimated); Last update posted 2013-06-11 (Estimated); Status verified 2013-06

CONDITIONS: Biomarkers of Stress in Emergency Physicians
Keywords: Stress, occupation, biomarkers, emergency, physicians
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Who Masked: Participant

ARMS (1):
- biomarkers of stress (Other): Comparison of biomarkers of stress in emergency physicians working a 24-hour shift or a 14-hour night shift
  Interventions: Behavioral: Comparison of biomarkers of stress

INTERVENTIONS:
Behavioral: Comparison of biomarkers of stress

SUMMARY:
A stressful state can lead to symptoms of mental exhaustion, physical fatigue, medical errors, and also increase coronary heart disease. Emergency physicians subjectively complain of stress related to changes in work shifts. Several potential biomarkers of stress have been described, but never investigated in emergency physician, who may represent a good model of stress due to the complex interplay between stress (life-and-death emergencies, which is the defining characteristic of their job), lack of sleep and fatigue due to repeated changes in shifts.The aim of this study was to compare biomarkers in emergency physicians working a 24-hour shift (24hS) or a 14-hour night shift (14hS), and in those working a control day (clerical work on return from leave). We also followed these markers three days following each shift (D3/24hS and D3/14hS).

DETAILED DESCRIPTION:
A stressful state can lead to symptoms of mental exhaustion and physical fatigue, detachment from work, and feelings of diminished competence. One of the health consequences of chronic stress at work is an increased risk of coronary heart disease. Emergency physicians subjectively complain of stress related to changes in work shifts. In occupational medicine, no marker of stress or fatigue has achieved consensus. Several potential biomarkers of stress have been described, but never investigated in emergency physician, who may represent a good model of stress due to the complex interplay between stress (life-and-death emergencies, which is the defining characteristic of their job), lack of sleep and fatigue due to repeated changes in shifts.The aim of this study was to compare HRV in emergency physicians working a 24-hour shift (24hS) or a 14-hour night shift (14hS), and in those working a control day (clerical work on return from leave). We will also follow these markers three days following each shift (D3/24hS and D3/14hS).

The psychological consequences of shifts will be assessed in terms of perceived stress and fatigue using visual analog scales. Potential biomarkers will be assessed through urine and saliva collections. Heart rate variability will be measured using 5-lead electrocardiogram. Psychological questionnaires will be completed only once during the control day. The workload during each shift will be estimated by: the total number of entries, the number of admissions, the number of outpatients (collected by computer), and the number of life-and- death emergencies (given by the emergency physician). Sleep duration, including naps, will be assessed by questionnaire (bed time - wake time) on the three-day tracking of each shift and on the control day.

Shift randomization: Latin squares were used to randomize the pattern of shifts and control day (24hS then 14hS then control day or any other combination).

Gaussian distribution of the data wil be tested by the Kolmogorov-Smirnov test. Data will be presented as mean ± standard deviation (SD). Comparisons between shifts will be made with ANOVA. Relationships between data will be assessed by Pearson correlation. Significance will be accepted at the p<0.05 level. Statistical procedures will be performed using SPSS Advanced Statistics software (SPSS Inc., Chicago, IL).

ELIGIBILITY:
Inclusion Criteria:

* emergency physician

Exclusion Criteria:

* endocrine disease, pregnancy, recent extraprofessional deleterious life event (such as death of a near relative, divorce), any current illness, drugs used to modulate inflammatory diseases (corticosteroids, anti-inflammatory drugs, immunomodulatory drugs), or any drugs with a chronotropic effect taken over the previous six months (beta blockers, diltiazem, verapamil, anxiolytics or antidepressants).

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-04; Primary Completion 2010-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Putative biomarkers of stress include heart rate variability (urinary and salivary steroids, saliva immunogobulin A, ...) | at day 1
  These biomarkers will be collected in emergency physicians

SECONDARY OUTCOMES:
perceived stress measured using visual analog scale (VAS) | at day 1
perceived fatigue (VAS) | at day 1
sleep duration (hours) | at day 1
sleep quality (VAS) | at ady 1
workload within the emergency department during the shifts | at day 1

CONTACTS AND LOCATIONS:
Overall Officials: Alain CHAMOUX, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- CHU Clermont-Ferrand, Clermont-Ferrand, France

REFERENCES:
- [Derived] Dutheil F, Marhar F, Boudet G, Perrier C, Naughton G, Chamoux A, Huguet P, Mermillod M, Saadaoui F, Moustafa F, Schmidt J. Maximal tachycardia and high cardiac strain during night shifts of emergency physicians. Int Arch Occup Environ Health. 2017 Aug;90(6):467-480. doi: 10.1007/s00420-017-1211-5. Epub 2017 Mar 7. PMID 28271382